CLINICAL TRIAL: NCT03339817
Title: Description Des Troubles Respiratoires Chez Les Patients Suivis Pour Une Sclérose en Plaques (SEP) sévère
Acronym: RespiMuS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C16-111; 2017-A01845-48 (Registry Identifier: RCB)
Record Dates: First submitted 2017-10-31; First posted 2017-11-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis; Respiration Disorders
MeSH Terms: conditions — Multiple Sclerosis; Respiration Disorders | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with severe MS (Other): polysomnography and functional pulmonary testings.
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — During polysomnographia and functional pulmonary testing, signs of diaphragmatic dysfunction responsible for respiratory disorders will be searched.
  Other Names: functional pulmonary testings

SUMMARY:
The purpose of this study is to describe respiratory disorders in patients with severe multiple sclerosis (EDSS from 6.5).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis criteria of multiple sclerosis (MS) fulfilling revised McDonald criteria (2010)
* EDSS score from 6.5
* no relapse during the 3 last months
* Informed consent prior to any study procedure

Exclusion Criteria:

* Any severe Chronic Obstructive Pulmonary Disease (III or IV)
* Pregnancy or woman with childbearing potential
* contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Polysomnography | Baseline only_during one night
  presence of phasic activation of respiratory muscles

SECONDARY OUTCOMES:
Respiratory function testing | Baseline only
  difference between vital capacity upright and supine position (liter)
Respiratory function testing | Baseline only
  maximal inspiratory pressure (mmHg)
Respiratory function testing | Baseline only
  maximal expiratory pressure (mmHg)
Respiratory function testing | Baseline only
  SNIP (mmHg)
Respiratory function testing | Baseline only
  peak flow (liter)
Cerebral and cervical spine MRI | Baseline only
  cerebral : 3DT1MPRAGE, T2 FLAIR, DWI / spine: 3DT1MPRAGE, axial T2 MEDIC, T2-WSPACE
Expanded Disability Status Scale (EDSS) | Baseline only
  Neurological assessment of disability related to multiple sclerosis, total score from 0 to 10
BICAMS | Baseline only
  Brief International Assessment for Multiple Sclerosis

CONTACTS AND LOCATIONS:
Overall Officials: Maillart Elisabeth, MD, Principal Investigator — Hopital de la Pitié Salpétrière
Locations (1):
- Département de Neurologie-Groupe Hospitalier Pitié-Salpêtrière, Paris, Paris, France

REFERENCES:
- [Result] Zeidan S, Redolfi S, Papeix C, Bodini B, Louapre C, Arnulf I, Maillart E. Unexpected REM sleep excess associated with a pontine lesion in multiple sclerosis. J Clin Sleep Med. 2021 May 1;17(5):1117-1119. doi: 10.5664/jcsm.9114. PMID 33538688